CLINICAL TRIAL: NCT06478758
Title: Ibuprofen Use on Post-operative Pain Following Cholecystectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAEK-230
Record Dates: First submitted 2024-06-12; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Acute Post-operative Pain
Keywords: intravenous ibuprofen; acetaminophen; laparoscopic cholecystectomy; postoperative pain control; analgesia; anti-inflammatory agents
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: The present study included ASA grade I-II participants aged 18-65 years scheduled for laparoscopic cholecystectomy. Participants with a history of allergies or hypersensitivity to the aforementioned agents, renal, hepatic or gastrointestinal disease, significant cognitive impairment, recent use of long-term nonsteroid anti-inflammatory and opioids, oral anticoagulant use or known bleeding disorders, diabetes or any other neuropathic diseases and those who were pregnant or breastfeeding were excluded from the study.
Who Masked: Investigator
Masking Description: Randomization of the participants was performed according to computer-generated random number tables, and allocation to a treatment group was performed using the envelope technique. For each participant taken the operating theater for laparoscopic cholecystectomy, an envelope was randomly selected and the code was recorded. The participants were unaware of which drug was being administered. The researcher who recorded the participants' demographic and follow-up data was also unaware of the type of drug being administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen group (Active Comparator): The acetaminophen group (n=35) received 1000 of mg acetaminophen intravenously in 100 mL saline at the end of the cholecystectomy.
  Interventions: Drug: Acetaminophen 100 MG/ML
- Ibuprofen group (Experimental): The ibuprofen group (n=36) was administered 800 mg of ibuprofen at the end of the cholecystectomy.
  Interventions: Drug: Ibuprofen 400 mg

INTERVENTIONS:
Drug: Ibuprofen 400 mg — The ibuprofen group (n=36) was administered 800 mg of ibuprofen . All procedures were performed with the same team. During surgery, a 20% increase in the participant's heart rate and mean arterial pressure remifentanil infusion was administered. During the postoperative period, all participants continued to receive acetaminophen at 8-hour intervals, and tramadol was given to those with a visual analog score above 4. In the recovery room, the participants with a visual analog score of > 4 were administered 100 mg of tramadol. All participants were prescribed acetaminophen every 8 hours postoperatively in whilst on the ward. Participants with a visual analog score of > 4 received rescue analgesia with 100 mg of tramadol. Visual analog score and vital parameters were recorded at 1, 2, 6, 12 and 24 h postoperatively. The incidence of nausea and vomiting during the 24 h postoperative period was also recorded.
  Arms: Ibuprofen group
Drug: Acetaminophen 100 MG/ML — The investigators administered 1000 mg of acetaminophen to the participants in Group A. A 20% increase in the participant's heart rate and mean arterial pressure was evaluated as pain and remifentanil infusion was administered. All participants continued to receive the routine application of acetaminophen at 8-hour intervals, and tramadol was given to those with a visual analog score above 4, postoperatively.In the recovery room, participants with a visual analog score of > 4 were administered 100 mg of tramadol. All participants were prescribed acetaminophen every 8 hours postoperatively in whilst on the ward. Participants with a visual analog score of > 4 received rescue analgesia with 100 mg of tramadol. Visual analog score and vital parameters were recorded at 1, 2, 6, 12 and 24 h postoperatively. The incidence of nausea and vomiting during the 24 h postoperative period was also recorded.
  Arms: Acetaminophen group

SUMMARY:
In this study, the investigators compared the effects of IV forms of ibuprofen and acetaminophen on pain perception and opioid consumption following laparoscopic cholecystectomy. Participants in Group I (group ibuprofen, n=35) were administered 800 mg of IV ibuprofen; participants in Group A (group acetaminophen, n=36) were administered 1000 mg of IV acetaminophen.

DETAILED DESCRIPTION:
Ibuprofen is a widely used NSAID that has antipyretic, analgesic, and anti-inflammatory effects. In this study, the investigators compared the effects of IV forms of ibuprofen and acetaminophen on pain perception and opioid consumption following laparoscopic cholecystectomy.The participants in this study were randomized into two groups. Participants in Group I (group ibuprofen, n=35) were administered 800 mg of IV ibuprofen; participants in Group A (group acetaminophen, n=36) were administered 1000 mg of IV acetaminophen. The investigators recorded demographic data including gender, age, ASA, BMI, duration of anesthesia and surgery, poNV, LOS, VAS scores and opioid consumption postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA grade I-II patients
* Aged 18-65 years

Exclusion Criteria:

* History of allergies or hypersensitivity to the aforementioned agents
* Renal, hepatic or gastrointestinal disease
* Significant cognitive impairment
* Recent use of long-term nonsteroid anti-inflammatory and opioids
* Oral anticoagulant use or known bleeding disorders
* Diabetes or any other neuropathic diseases
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
VAS scores in the postoperative period | 24 hour
  Primary outcome was to reduce the VAS scores in the postoperative period. For this purpose the investigators recorded VAS scores at the 1, 2, 6, 12 and 24 h postoperatively.

SECONDARY OUTCOMES:
Opioid consumption and length of stay | 24 hour
  Secondary outcome was any decrease in opioid consumption and hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Azime Bulut, MD, Principal Investigator — Giresun University
Locations (1):
- Giresun University, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ahiskalioglu EO, Ahiskalioglu A, Aydin P, Yayik AM, Temiz A. Effects of single-dose preemptive intravenous ibuprofen on postoperative opioid consumption and acute pain after laparoscopic cholecystectomy. Medicine (Baltimore). 2017 Feb;96(8):e6200. doi: 10.1097/MD.0000000000006200. PMID 28225506
- [Result] Ciftci B, Ekinci M, Celik EC, Kaciroglu A, Karakaya MA, Demiraran Y, Ozdenkaya Y. Comparison of Intravenous Ibuprofen and Paracetamol for Postoperative Pain Management after Laparoscopic Sleeve Gastrectomy. A Randomized Controlled Study. Obes Surg. 2019 Mar;29(3):765-770. doi: 10.1007/s11695-018-3613-1. PMID 30474791
- [Result] Mohammadian Erdi A, Arabzadeh A, Isazadehfar K, Masoumzadeh M, Bahadoram M. Comparing the Efficacy and Side Effects of Intravenous Ibuprofen and Acetaminophen in Pain Control Following Laparoscopic Cholecystectomy. World J Plast Surg. 2022 Mar;11(1):117-124. doi: 10.52547/wjps.11.1.117. PMID 35592235
- [Result] Celik EC, Kara D, Koc E, Yayik AM. The comparison of single-dose preemptive intravenous ibuprofen and paracetamol on postoperative pain scores and opioid consumption after open septorhinoplasty: a randomized controlled study. Eur Arch Otorhinolaryngol. 2018 Sep;275(9):2259-2263. doi: 10.1007/s00405-018-5065-6. Epub 2018 Jul 18. PMID 30022362